CLINICAL TRIAL: NCT05651477
Title: Establishing a Sub Cohort for Relationship Between Health Risk and Occupational Exposure of Emergency Medical Workers
Brief Title: Relationship Between Health Risk and Occupational Exposure of ED
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-09-044-001
Record Dates: First submitted 2022-10-30; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-10

CONDITIONS: Occupational Exposure; Occupational Problems; Occupational Burnout; Medical Emergencies
Keywords: Wearable Device; Smart Watch; Internet of Things; IoT; Personal Health Record; PHR
MeSH Terms: conditions — Burnout, Professional | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doctor: Doctors of the Emergency department conduct questionnaires about occupational, mental, physical factors on their health.
  Interventions: Device: Wearable Device (Smart Watch); Device: Edge-Box
- Nurses: Nurses of the Emergency department conduct questionnaires about occupational, mental, physical factors on their health.
  Interventions: Device: Wearable Device (Smart Watch); Device: Edge-Box

INTERVENTIONS:
Device: Wearable Device (Smart Watch) — A smart watch refers to an embedded system portable watch equipped with improved functions than a general watch, and is almost always in the form of a wrist watch. The device we are using is the Samsung Galaxy 4 (SM-R860/870).
Device: Edge-Box — Edge-Box collects data such as air. The device we are using is the TDS Mfepc-4C2R.

SUMMARY:
This study established a sub-cohort of emergency medical workers, for the development of health care and disease prevention solution, by identifying epidemiological characteristics and factors related to occupational exposure. Each life-log or environment-log data will be collected by wearable device (e.g. smart-watch) and IoT (e.g. Edge-box). From collected data, relationship between health risks and occupational exposure of emergency medical workers will be determined.

DETAILED DESCRIPTION:
Background : In South Korea, incidence of medical emergency is increasing, and 10 million people are using emergency medical services annually. Emergency medical services, which are directly related to the lives of the people, are essential, but medical staffs engaged in the department are reported to be at high risk due to health-related problems and poor working conditions. Although their general health status is confirmed through periodical health screening, there is a lack of research regarding each really individual health problems.

Objective : This study aims to establish a sub-cohort research system of emergency medical workers to develop disease prevention and health management solutions by identifying relationship between health risk and occupational exposure.

Design : Prospective Observational Cohort Study

Setting : In the Department of Emergency in 5 medical institutions

Enrollment : To be recruited by invitation from the prior cohort (NCT04883684) that consist of 105 doctors or nurses

Data Collection-1 : Life-log data collection by wearable device (smart watch) Participants wear smart watch freely during 12 months. Participants are recommended to wear a watch for at least 10 hours or more a day, and informed it must be worn during work and sleep, while this study assumes wearing a watch without any special intervention in daily life. Participants should access the watch app to transmit the saved data in watch, 2 times a week (Monday and Thursday)

Data Collection-2 : Environment-log data collection by edge-box (TDS Mfepc-4C2R) Among the five institutions where the participants works, Samsung Medical Center collects and manages data by installing 4 edge boxes in emergency medical centers to measure air quality.

ELIGIBILITY:
Inclusion Criteria:

* An Emergency Medical Worker (doctor, nurse) subject recruited from prior cohort construction studies.
* An adult aged 18 or older, who voluntarily agrees and signs.
* A subject who has not experienced occupational disease or damage within four weeks from the time of establishing a sub-cohort.

Exclusion Criteria:

* An subject who was recruited from prior cohort construction studies, but withdraws the agrees at the time of establishing a sub-cohort
* A subject who does not agree to participate in this study or withdraw the consent after agreement.
* A subject who is not engaged in work, such as leave of absence.
* A subject who has experienced occupational disease or damage within four weeks from the time of establishing a sub-cohort.
* A subject who is legally unable to participate in clinical research or unable to participate in clinical research at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical workers of the emergency department in the tertiary hospitals in Korea
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Some Change Value of Life-log during the Specific Interval | To access the watch app to transmit the saved data in watch, 2 times a week (Monday and Thursday). There is no specific event, but the time frame is transmitted throughout the study period (December 31, 2023).
  Life-log means a record of an individual's daily life. Participants are recommended to wear a watch for at least 10 hours or more a day during work and sleep, while wearing a watch without any special intervention in daily life.
Some Change Value of Environment-log during the Specific Interval | To transmit the saved data in box, automatically every day. There is no specific event, but the time frame is transmitted throughout the study period (December 31, 2023)
  Environment-log means a continuous record of a working space, and it mainly measures the air quality.

CONTACTS AND LOCATIONS:
Overall Officials: Taerim Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
This is a multicentered study and there are researchers of other institutes, therefore, IPD can be available to them.